CLINICAL TRIAL: NCT04792047
Title: Increased Pericoronary Fat Attenuation Index is Associated With High-risk Plaque and Local Immune-inflammatory Activation in Patients With Non-ST Elevation Acute Coronary Syndrome
Brief Title: Pericoronary Fat Attenuation Index and High-risk Plaque in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FAI and HRP study
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Acute Coronary Syndrome
Keywords: pericoronary fat attenuation index; high-risk plaque
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lesions with perivasular FAI greater than ≥-70.1
  Interventions: Diagnostic Test: HRP frequency, plaque compostion and local immune-inflammatory activation
- Lesions with perivasular FAI greater than <-70.1
  Interventions: Diagnostic Test: HRP frequency, plaque compostion and local immune-inflammatory activation

INTERVENTIONS:
Diagnostic Test: HRP frequency, plaque compostion and local immune-inflammatory activation — HRP frequency, plaque compostion were detected by CCTA method. Local T cell subsets and their intracellular cytokines levels were detected by Flow Cytometry.

SUMMARY:
This study aimed to investigate the relationship between CCTA-based pericoronary inflammation and plaque features as well as local immune-inflammatory biomarkers in ACS patients. It is hypothesized that perivascular FAI might serve as a reliable sensor of coronary immune-inflammatory disorder, and closely related to the plaque vulnerability.

DETAILED DESCRIPTION:
The pericoronary fat attenuation index (FAI), which capture by standard coronary computed tomography angiography (CCTA), has emerged as a novel imaging biomarker of coronary inflammation. This study aimed to assess whether increased Pericoronary FAI on CCTA are associated with high-risk plaque (HRP) feature as well as local T cell subsets and their intracellular cytokines levels in non-ST elevation acute coronary syndromes ( ACS) patients. 195 lesions in 130 non-ST elevation ACS patients were prospectively enrolled and evaluated by CCTA and coronary angiography in this study. Blood were taken from coronary artery immediately after the diagnostic angiogram. Local T cell subsets and their intracellular cytokines levels were detected by Flow Cytometry. CCTA and pericoronary FAI examinations were performed using a 320-detecor (Aquilion ONE, Toshiba Medical Systems, Otawara, Japan) Systems. Coronary plaque characteristics were analyzed cross each of the main coronary arteries using commercialized software package (Qangio CT, Medis, The Netherlands).

ELIGIBILITY:
Inclusion Criteria:

* non-ST-elevation ACS (non-ST-elevation myocardial infarction or unstable angina) age from 18 to 75 years which underwent CCTA were prospectively enrolled in this study.

Exclusion Criteria:

1. Patients needed an immediate (<2 h) or early invasive strategy (<24 h) according to guidelines were excluded: including those presented with haemodynamic instability or cardiogenic shock, life-threatening arrhythmia or cardiac arrest, mechanical complication, acute heart failure, dynamic ST or T wave changes, GRACE score >140;
2. Subjects with previous history of coronary artery bypass graft surgery or PCI, immune system disorder, tumor, acute/chronic infection, atrial fibrillation, end-stage renal failure, iodine-containing contrast allergy were also excluded.
3. After CCTA performance, we also exclude patients with no significant (≥50%) stenosis on major epicardial vessels and those refused subsequent angiography.
4. Participants with total obstruction on major epicardial vessel, or insufficient image quality for FAI and QangioCT analysis, as well as lack of blood sample were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2019 and January 2020, a total of 130 patients with 195 lesions were included in our study for final analysis.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency of HRP by CCTA | coronary CTA analysis, before angiography
  HRP features were defined according to previous studies as follow: low-attenuation plaque (LAP), mean CT number <30 HU; positive remodeling(PR), remodeling index, >1.1; spotty calcification(SC), intraplaque calcification ≤3 mm; Napkin-ring sign, low intraplaque attenuation surrounded by a higher attenuation rim.

SECONDARY OUTCOMES:
Distribution of plaque composition by Qangio | coronary CTA analysis, before angiography
  HU -30 to 75, for necrotic core;HU 76-130 for fibro-fatty; HU131-350 for fibrous, and HU> 351 for dense calcium.

OTHER OUTCOMES:
Concentration of local immune-inflammatory cytokines | blood were taken immediately after the diagnostic angiography
  quantification of local immune-inflammatory cytokines
Concentration of local T subset | blood were taken immediately after the diagnostic angiography
  quantification of local T subset

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, Principal Investigator — RenJi Hospital
Locations (1):
- Cardiology, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun JT, Sheng XC, Feng Q, Yin Y, Li Z, Ding S, Pu J. Pericoronary Fat Attenuation Index Is Associated With Vulnerable Plaque Components and Local Immune-Inflammatory Activation in Patients With Non-ST Elevation Acute Coronary Syndrome. J Am Heart Assoc. 2022 Jan 18;11(2):e022879. doi: 10.1161/JAHA.121.022879. Epub 2022 Jan 13. PMID 35023363